CLINICAL TRIAL: NCT03226912
Title: The PREDICT Study- a Registry in Critically Ill Patients to Determine Predictors of Disability Free Survival
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Other Study IDs: ANZIC-RC/CH002
Record Dates: First submitted 2017-07-17; First posted 2017-07-24 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Critical Illness; Mechanical Ventilation Complication; Disabilities Multiple; Quality of Life; Physical Disability; Anxiety; Depression; Cognitive Change
MeSH Terms: conditions — Critical Illness; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As mortality from critical illness has reduced, the importance of measuring disabilities (cognitive, functional and psychological) in surviving critically ill patients has become more important. Currently, the causes, long-term effects and frequency of disabilities in patients surviving ICU in Australia are unknown. In the US and UK, studies have been undertaken to assess the effects of specific long-term outcomes, such as functional disability and depression, which found long-term disabilities were much higher than baselines (pre-illness function) and ongoing at five years after ICU discharge. In order to improve quality of life of ICU survivors and ensure that medical specialists apply appropriate interventions to reduce the cost of these surviving patients on the community, the PREDICT management committee proposes the introduction of a patient-reported outcomes registry.

DETAILED DESCRIPTION:
Critical illness affects more than 100,000 patients per year in Australia and more than 25,000 per year in Victoria. Although, hospital mortality in Australia and New Zealand has decreased over the past decade in all major admission categories, and 90% of these patients now survive to return to live in the community, just 28% of previously working ICU survivors are currently expected to return to work after discharge. Most ICU survivors suffer from post-ICU accelerated neurocognitive decline, prolonged neuromuscular weakness, post-traumatic stress disorder, depression, and/or anxiety. The recovery process and long-term outcomes for critically ill patients may be poor, and they can be improved by appropriate interventions, continual support and tracking of patients post-ICU as they recover, as opposed to being discharged to a single general practitioner who may not have the resources to provide adequate rehabilitation. Although this method has been previously seen as cost-effective, this approach actually carries huge costs for the community of the individuals as they often cannot return to work and have ultimately lost independence. By assessing risk factors and measuring long-term outcomes of patient's post-ICU, the severity of the community burden could be decreased with the application of suitable interventions.

The PREDICT study follows on from the successful completion of the ICU-Recovery Project (HREC Reference Alfred Health 180/14) which found that disability was prevalent in ICU and was associated with sepsis and pre-existing mental health problems. The PREDICT study will measure disability-free survival, psychological function, cognitive function and quality of life with health economic outcomes in critically ill patients 3 and 6 months after ICU admission. The study will confirm the predictors of disability-free survival.

These patients add to the community burden and also influence community and rehabilitation costs. Our aim is to improve long-term patient outcomes through: improving sedation practices, delirium prevention, neurocognitive stimulation, early mobilisation, post-ICU follow-up, and functional and psychological rehabilitation. This study is required for the evaluation of hospital and post-ICU rehabilitation practice as there is insufficient evidence to alter current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients who have been mechanically ventilated for over 24 hours
* Patients 18 years or older

Exclusion Criteria:

* A Proven or suspected acute primary brain process that is likely to result in global impairment of conscious level or cognition (e.g. TBI, SAH, stroke or hypoxic brain injury after cardiac arrest)
* Second or subsequent admission to ICU during a single hospital admission
* Participants who do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 critically ill patients who were mechanically ventilated > 24 hours in an intensive care unit who have survived to hospital discharge.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Development of a risk-prediction model for disability-free survival in high risk patients (after > 24 hours of mechanical ventilation) | 3-6 months post ICU admission
  Development of a risk-prediction model for disability-free survival in high risk patients (after > 24 hours of mechanical ventilation)

SECONDARY OUTCOMES:
Health related quality of life (HRQOL) | 3-6 months post ICU admission
  Health related quality of life (HRQOL) measured with EQ5D before ICU
Pre ICU health status | 3 months post ICU admission
  pre ICU health status measured by retrospective EQ5D
Global function | 3-6 months post ICU admission
  Global function measured with the WHODAS
Physical activity at 6 months | 6 months post ICU admission
  Physical activity at 6 months measured with the IADL
Cognitive function at 6 months | 6 months post ICU admission
  Cognetive function measured using the MOCA blind
Anxiety and depression at 6 months will be assessed | 6 months post ICU admission
  Anxiety and depression at 6 months will be assessed with the Hospital Anxiety and Depression Scale (HADS) and the Impact of Event Scale (IES-R)
Return to work at 3 and 6 months | 3-6 months post ICU admission
  Return to work at 3 and 6 months will be measured using extra questions
Pre ICU disability and work status | 3 months post ICU admission
  Pre ICU disability and work status measured using the WHODAS

CONTACTS AND LOCATIONS:
Locations (1):
- Australian New Zealand Intensive Care Reseearch Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Higgins AM, Neto AS, Bailey M, Barrett J, Bellomo R, Cooper DJ, Gabbe BJ, Linke N, Myles PS, Paton M, Philpot S, Shulman M, Young M, Hodgson CL; PREDICT Study Investigators. Predictors of death and new disability after critical illness: a multicentre prospective cohort study. Intensive Care Med. 2021 Jul;47(7):772-781. doi: 10.1007/s00134-021-06438-7. Epub 2021 Jun 5. PMID 34089063
- [Derived] Hodgson CL, Higgins AM, Bailey M, Barrett J, Bellomo R, Cooper DJ, Gabbe BJ, Iwashyna T, Linke N, Myles PS, Paton M, Philpot S, Shulman M, Young M, Serpa Neto A; PREDICT Study Investigators. Comparison of 6-month outcomes of sepsis versus non-sepsis critically ill patients receiving mechanical ventilation. Crit Care. 2022 Jun 13;26(1):174. doi: 10.1186/s13054-022-04041-w. PMID 35698201